CLINICAL TRIAL: NCT06439888
Title: Pan-lesions SBRT Combined With Lymphocyte Support Through ATRA-driven Blockade of MDSC in Patients With Oligo-metastatic Solid Cancer
Brief Title: Lymphocyte Support to SBRT in Patients With Oligo-metastatic Solid Cancer
Acronym: LySATRA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-500680-13-00; 2022/3511 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Oligometastatic Disease; Solid Tumor, Adult
MeSH Terms: interventions — Tretinoin; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part I : Stereotactic Body Radiation Therapy + All-trans retinoic acid (Experimental): Part I will allow to evaluate the safety of pan-metastases directed SBRT combined with ATRA in N=6 patients.
  * SBRT to all lesions more than 1.5cm, on Monday up to Friday, over a maximum of 2 weeks,
  * ATRA 150 mg/m2/day given orally for 3 days every 3 weeks for a maximum of 4 cycles (about 3 months), starting on the same day as SBRT.
  Interventions: Drug: all-trans retinoic acid; Radiation: Stereotactic Body Radiation Therapy
- Part II : Stereotactic Body Radiation Therapy + All-trans retinoic acid (Experimental): Part II will allow to evaluate the lympho-protective efficacy of ATRA upon radiation-induced lymphopenia. The experimental arm consists in :
  * SBRT to all lesions more than 1.5cm, on Monday up to Friday, over a maximum of 2 weeks,
  * ATRA 150 mg/m2/day given orally for 3 days every 3 weeks for a maximum of 4 cycles (about 3 months), starting on the same day as SBRT.
  Interventions: Drug: all-trans retinoic acid; Radiation: Stereotactic Body Radiation Therapy
- Part II : Stereotactic Body Radiation Therapy alone (Placebo Comparator): Part II will allow to evaluate the lympho-protective efficacy of ATRA upon radiation-induced lymphopenia. The control arm consists in :
  - SBRT to all lesions more than 1.5cm, on Monday up to Friday, over a maximum of 2 weeks
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: all-trans retinoic acid — per os treatment, started from the same day as SBRT, during 3 successive days, every 3 weeks, for a maximum of 4 cycles
  Other Names: Tretinoin; VESANOID
  Arms: Part I : Stereotactic Body Radiation Therapy + All-trans retinoic acid; Part II : Stereotactic Body Radiation Therapy + All-trans retinoic acid
Radiation: Stereotactic Body Radiation Therapy — Standard of Care, planned over 1 or 2 weeks, every lesions must be irradiated

SUMMARY:
The goal of this clinical trial is to assess safety of pan-metastases directed SBRT combined with ATRA and the lympho-protective efficacy of ATRA upon radiation-induced lymphopenia.

This is a French bicentric, open label, phase I/II clinical study that will comprise two parts. Part I will evaluate the safety of the combination based on a single-arm safety run design, while Part II will be randomized (ratio 1:1) and will study SBRT with or without ATRA.

Patients enrolled will be treated with:

* SBRT to all lesions more than 1cm, on week days (from Monday to Friday), over a maximum of 2 weeks,
* With or without (for part II patients randomized in the control arm) ATRA therapy: ATRA 150 mg/m^2/day for 3 days every 3 weeks for a maximum of 4 cycles (about 3 months), starting on the first day of radiation therapy.

The expected rate of patients who will have lymphopenia of grade 2 or higher in the control arm at 6 weeks post-radiotherapy is 50%.

At a one-sided level of statistical significance of 0.07, the randomization of 52 patients (26 patients in each arm) will provide 85% power to detect a decrease in this rate to 15% in the SBRT+ATRA arm, using Fisher's exact test.

DETAILED DESCRIPTION:
Ablative radiotherapy - also called stereotactic body radiation therapy (SBRT) - can achieve durable control of tumor lesions and appears as a highly promising strategy to extend overall survival of patients with oligo-metastatic diseases. Radiotherapy has recognized immunomodulatory effects: it triggers immunogenic cell death and reprogramming of the tumor immune microenvironment, which eventually results in a systemic antitumor response following focal radiation treatment. This is called the abscopal effect (distant out-of-the-field lesions that shrink after focal irradiation). Unfortunately, evidences show that this is directly counteracted by the toxic effects of radiotherapy on cytotoxic lymphocytes, which are highly radiosensitive.

Recent data support the fact that radiation-induced lymphopenia is mostly driven by the deregulation of the myeloid-lymphoid imbalance following radiation therapy, with aberrant myelopoiesis and high levels of tumor infiltration by myeloid-derived suppressive cells (MDSC). In preclinical models, pharmacological blockade of MDSC combined with radiation therapy successfully abrogated radiation-induced lymphopenia and significantly improved survival outcomes.

All trans retinoic acid (ATRA, also known as tretinoin) is a vitamin A derivative that has a market authorization for the treatment of acute promyelocytic leukemia as it efficiently induces differentiation of abnormal promyelocytes. Similarly, several clinical studies report that ATRA can differentiate MDSCs into mature myeloid cells, with a positive effect on the count of activated cluster of differentiation 8 (CD8+) lymphocytes.

This clinical trial will provide the clinical proof-of-concept that adding ATRA to pan-metastases SBRT is safe in humans, prevents severe and prolonged lymphopenia and therefore, may foster a radiation-induced systemic anticancer immune response sufficient to increase survival in patients with cancer at the oligo-metastatic stage.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible for enrolment in the study only if ALL of the following criteria apply:

I1. Adult male or female patients (≥ 18 years of age at inclusion);

I2. Histologically or cytologically proven solid cancer at the oligometastatic stage and/or oligoprogressive amenable to pan-lesion SBRT, as defined by:

1. [1-5] active tumor lesions with a largest diameter comprised between [1-5] cm,
2. The disease can be either genuinely oligometastatic, oligoprogressive, or an induced oligometastatic disease
3. All active tumor lesions (progressive and/or hypermetabolic) that match criterion I2a must be eligible to SBRT in terms of location and radiotherapy constraints. 'Active lesion' is defined as either: hypermetabolic on PET-scan, recent increase of >20% of its largest diameter on CT-scan, and/or any new lesion of ≥ 1cm on the most recent CT-scan
4. SBRT to all active lesions must be feasible over a two-week period,
5. Whatever the primary tumor type I3. Patients must agree to comply with biopsy and blood sampling for research purpose;

I4. Minimal wash-out periods from last administration of treatments to the first day of SBRT must be:

1. Systemic chemotherapy including cytotoxic, immunotherapy, targeted therapy, hormone therapy, any investigational agent > 4 weeks,
2. Immunosuppressive medication > 4 weeks, with the exceptions of intranasal, topical, and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceeding 10 mg/day of prednisone, or an equivalent corticosteroid,
3. Live attenuated vaccination > 4 weeks,
4. Major surgery > 4 weeks; I5. WHO 0-1 and ECOG Performance Status 0-1;

I6. Patients must have adequate organ function defined as follows:

1. White blood cell count of ≥ 1,500/mm3,
2. Lymphocyte count of ≥ 800/mm3,
3. Platelet count of ≥ 100,000/mm3,
4. Hemoglobin > 9 g/dL, Serum ALT and AST ≤2.5 ULN (or if liver metastases are present must be ≤ 5x ULN)

f. Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance; I7. Female patients must either be of non-reproductive potential or must have a negative serum pregnancy test within 3 days prior to the initiation of the study drug and/or perform a urine test in addition to the serum test before the first dose of ATRA, if the result of the serum test cannot be obtained within 3 days. Fertile men with a female partner of childbearing potential must agree to use male condom plus spermicide and childbearing potential women must have agreed to use at least one highly effective contraceptive method during treatment on this trial and for up to 1 month after the last dose of ATRA; Pregnancy testing and contraception counseling should be repeated monthly throughout the period of ATRA treatment.

I8. Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol; I9. Patients must be affiliated to a social security system or beneficiary of the same 4.2. Non-inclusion criteria

Participants are not eligible for enrolment in the study if ANY of the following criteria applies:

E1. Evidence of disease rapidly progressing at the time of screening according to the two last best-fitted imaging modalities (CT-scans, MRI, PET-scan), at the discretion of the investigator and the multidisciplinary board (RCP); E2. Any evidence of brain metastasis; E3. Any situation where irradiation of the target site(s) would imply re-irradiation of a formerly irradiated tumor site; E4. Bone metastasis located in a femoral bone if risk of pending fracture is high; E5. Liver metastasis adjacent to the stomach or small bowel and liver metastasis that leads to a volume of uninvolved liver < 700 cc; E6. Patients with any concurrent severe condition (grade 3 or beyond according to CTCAE V5.0) and/or uncontrolled medical condition that could compromise participation in the study; E7. Any psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent; E8. Active secondary malignancy unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the Sponsor. Examples of the latter include basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, and isolated elevation of prostate-specific antigen. Patients with a completely treated prior malignancy who are no longer treated (including maintenance therapy) and no evidence of disease for ≥ 2 years are eligible; E9. Chronic treatment with systemic corticosteroids or another immunosuppressant including, but not limited to systemic corticosteroids at doses exceeding 10 mg/day of prednisone or equivalent, methotrexate, azathioprine, and TNF-α blockers. Use of immunosuppressive medications for the management of investigational product-related AEs or in subjects with contrast allergies is acceptable. The use of topical, inhaled and intranasal corticosteroids is permitted; E10. Patients with tumor(s) that invade major vessels, as shown unequivocally by imaging studies; E11. Patients with central lung metastasis (i.e within 2 cm from hilum) that are cavitary as shown unequivocally by imaging studies; E12. Persisting significant toxicities related to prior treatments i.e. ≥ Grade 2 adverse event according to CTCAE V5.0 criteria, except for alopecia and biological values defined in inclusion criteria I6; E13. Known allergy or hypersensitivity to the study drug. The study drug is contraindicated in patients with soy or peanut allergy; E14. Positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS); E15. Patients at risk of QT prolongation (including patients with hypokaliemia, baseline QT/QTc interval > 470 ms (for women) and > 450 ms (for men)); E16. Pregnant or breastfeeding women; E17. Persons deprived of their freedom or under guardianship, or for whom it would be impossible to undergo the medical follow-up required by the trial, for geographic, social or psychological reasons.

Women of childbearing potential must have a negative serum β-HCG pregnancy test within 3 days prior to the administration of the first study treatment (and/or a urine test).

Sexually active women of childbearing potential must agree to use a highly effective method of contraception, or to abstain from sexual activity during the study and for at least 1 months after the last study treatment administration.

Sexually active male patients must agree to use condom during the study and for at least 1 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception.

Of note:

A woman is considered of childbearing potential following menarche and until becoming post-menopausal (≥ 12 months of non-therapy-induced amenorrhea) unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral oophorectomy and bilateral salpingectomy.

A highly effective birth control method is a one which can achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include: combined (estrogen and progestogen containing) hormonal contraception; progestogen-only hormonal contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence during the entire period of risk associated with study treatment. To prevent the risk of interaction between the study drug and hormonal contraceptives, hormonal contraceptives should be supplemented with a barrier method (preferably male condom). Following methods are considered as unacceptable methods (non-exhaustive list): periodic abstinence (calendar, symptothermal, post-ovulation methods) and withdrawal (coitus interruptus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | from the first intake to 3 weeks after the treatment initiation
  Dose-limiting toxicity (DLT) is defined as an adverse event reported during the first three weeks of treatment that is possibly related to study intervention and fulfills any one of the DLT criteria using CTCAE Version 5.0
Lympho-protective efficacy | At 6 weeks after SBRT completion
  Rate of patients with lymphopenia grade 2 or higher at 6 weeks after treatment completion (as absolute lymphocyte count less than 800/mm3 (CTCAE V5.0))

SECONDARY OUTCOMES:
Control rates | from 6 weeks to 1 year after SBRT
  Control rates on the treated lesions
Objective response rate | from 6 weeks to 1 year after SBRT
  Objective response rate
Duration of response | from 6 weeks to 1 year after SBRT
  Duration of response
Progression-free survival | from 6 weeks to 1 year after SBRT
  Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Eric DEUTSCH, PhD, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (2):
- France (2):
  - Centre Léon Bérard, Lyon
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No